CLINICAL TRIAL: NCT01576978
Title: Hatha Yoga Exercises in Pelvic and Lumbar Back Pain in Pregnant Woman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Roseny Flávia Martins, principal investigator (student), University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: w7tgp7jt
Record Dates: First submitted 2012-02-24; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: LUMBAR BACK PAIN; PELVIC PAIN; PREGNANCY
Keywords: LUMBAR BACK pain; PELVIC PAIN; PREGNANCY; HATHA YOGA
MeSH Terms: conditions — Low Back Pain; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- postural orientations (Active Comparator): The group of postural orientations receive a pamphlet containing information about the sitting, standing and lying postures to be performed at home for 10 weeks.The marking of the note pain will be before and after 10 weeks.
  Interventions: Behavioral: hatha yoga
- hatha yoga exercises (Active Comparator): The allocates women will participate in the Hatha yoga class for 10 weeks. At first in class, the women will make a note of pain according to VAS. Class Moments: heating ten minutes, forty minutes postures of stretching and strengthening exercises and breathing exercises, ten minutes of relaxation and meditation. Marking note of pain after practice.
  Interventions: Behavioral: hatha yoga

INTERVENTIONS:
Behavioral: hatha yoga — The women's group of Yoga will participate in ten week sessions of Yoga once a week for an hour. The sessions will be taught by instructor of Hatha Yoga. For the intervention were chosen 37 postures, three breathing exercises. The sessions were divided into three stages: quieting the mind , breathing rate and the heating of the main joints, postures and breathing exercises, meditation and relaxation. At the beginning and end of each session, we evaluated the pain intensity.Pregnant women in the control group Postural orientations will receive a booklet containing guidelines postural figures and explanatory text on some possible changes in the curvatures of the spine during pregnancy suggestions for positioning of the spine for daily activities, lying postures, sitting and standing. After ten weeks the two groups will be scheduled for the final collection of data.

SUMMARY:
The aim of this study is to identify evaluate the effectiveness of stretching exercises of Hatha Yoga method in pregnant women with back pain and posterior pelvic City Paulínia. -There will be a randomized clinical trial with 60 pregnant women with these symptoms. They will be randomly divided into 2 groups. The group A will perform the exercises of Hatha Yoga for ten weeks, once a week group B postural follow the guidelines recommended for the treatment of these pains, for ten weeks. Will be used as a technique for evaluating the Visual Analogue Scale to measure pain intensity and confirmation tests of the lumbar and posterior pelvic pain in order to differentiate them. A descriptive statistical analysis of univariate and bivariate distributions will be made through frequency and graphical representation. The association between the variables will be tested by statistical tests: [chi-square (X ²)], Fisher's exact test, Student's t test or Mann-Whitney, [Student's t test to compare means], ANOVA for the analysis of effects between the groups. [The significance level is predetermined to 5%]. The data will be analyzed in EPI-INFO 2000. SAS 9.0 and from the database created .

DETAILED DESCRIPTION:
OBJECTIVES

General Purpose Identify the percentage of pregnant women with spinal postural pains in antenatal services in the city of Paulinia and evaluate the effectiveness of the Classical Yoga exercises for the lumbar and posterior pelvic pains in the group of women who will do the exercises, as well as developments pain intensity in patients with and without exercise.

Specific Objectives

* Identify the percentage of pregnant women with postural pains in the spine.
* Measure the intensity of pain and at the beginning and end of intervention in both groups.
* Measure the intensity of pain and at the beginning and end of each exercise session.
* To compare the evolution of pain - lower back and posterior pelvic pain - in the group with and without exercise.
* To compare the evolution of pain - lower back and posterior pelvic pain - in the group with Yoga exercises.

ASSUMPTIONS

* Half of pregnant women report symptoms of postural pains in the spine.
* A significantly higher percentage of pregnant women who will do the Yoga exercises during pregnancy report improvement in pain intensity - low back and / or posterior pelvic pain - compared with the control group.
* A significantly higher percentage of pregnant women present pain intensity increased at the beginning compared to the end of the session.
* A significantly higher percentage of pregnant women report a decrease in intensity of back pain and posterior pelvic pain when compared to the control group.
* A significantly higher percentage of pregnant women report improvement in low back pain over the posterior pelvic pain in the group with Yoga exercises.

SUBJECTS AND METHODS:

Design Identification of the percentage of pregnant women with postural pains in the spine in health units and clinical trial, prospective, randomized and controlled.

Sample Size To calculate the sample size was calculated as the average change in pain intensity referred to the global active stretching group at the end of the first and eighth week of treatment. The mean and standard deviation of the intensity of pain at the end of the first week was 4.88 SD 3.056 and at the end of the eighth week 0.85 SD 1.875 (Martins & PINTO E SILVA, 2005 b) The assumption is that the effect of treatment with yoga is similar to that found with the global active stretching.

Considering a significance level of 5%, a test power of 80%, based on the mean difference reported and adopting the paired t-test, the smallest sample size required is n = 7 women in each group.

However, for purposes of research and publication is suggested to adopt an "n" greater than 30 women per group.

ELIGIBILITY:
Inclusion Criteria:

* Lower back pain and / or posterior pelvic pain when completing the interview. Gestational age greater than or equal to 12 weeks.

Exclusion Criteria:

* Twin pregnancy. Medical restrictions on the exercise. Be doing physical therapy for the symptom of back pain and / or posterior pelvic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale (VAS) | 10 weeks
  Ratings of pain intensity according to the pregnant woman. Checking the initial interview, the beginning and end of each session of Yoga. The scale will be presented to the patient with a drawing where you see three little faces on a graphic scale, rating pain in ascending order, with a score of zero to ten (Olsen, NOLAN, Kori, 1992)
confirmatory low back pain test | 10 weeks
  The therapist will ask the mother to stand with feet together, the woman held the bending bending the trunk forward until the time you start bending the legs. It is positive if patient reported back pain and reported pain with palpation of the musculature of this area and in moving the trunk in a circle.
Confirmatory pelvic pain test | 10 weeks
  The therapist will place the pregnant woman lying supine, ask for a leg flexion and extension of the other on the floor. The femoral leg will be bent in the vertical and the physiotherapist push towards the ground, simultaneously stabilizing the pelvis. It is positive when the patient to recognize the pain .Low back pain, Trunk Flexion the therapist will ask the mother to stand with feet together, the woman held the bending bending the trunk forward until the time you start bending the legs. It is positive if patient reported pain in the deep gluteal area and turnning night on the bed.

CONTACTS AND LOCATIONS:
Overall Officials: Roseny F Martins, Msc, Principal Investigator — Universtity of Campinas

REFERENCES:
- [Derived] Martins RF, Pinto e Silva JL. Treatment of pregnancy-related lumbar and pelvic girdle pain by the yoga method: a randomized controlled study. J Altern Complement Med. 2014 Jan;20(1):24-31. doi: 10.1089/acm.2012.0715. Epub 2013 Mar 18. PMID 23506189